CLINICAL TRIAL: NCT04512885
Title: Study of the Acceptability of a New Distance-learning Tool for Functional Insulin Therapy "MyFIT" by Patients With Type 1 Diabetes (T1D) and by Healthcare Professionals
Brief Title: Study of Acceptability of a New Distance-learning Tool "MyFIT"
Acronym: MyFIT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, EVA FEIGERLOVA, Assistant Professor of Endocrinology, Central Hospital, Nancy, France
Other Study IDs: 2020PI162-49
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 1 diabetes
  Interventions: Other: Survey
- Health professionals
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey via questionnaire

SUMMARY:
The investigators developed an on-line learning tool "MyFIT" enabling to patients with T1D to acquire the knowledge and skills for practicing functional insulin therapy from their home.

The aim of the present study is to evaluate the acceptability of this new learning modality via the tool "MyFIT" by the patients and by the health professionnals.

ELIGIBILITY:
Inclusion Criteria:

* type one diabetes on intensified insulin therapy

Exclusion Criteria:

* Hearing loss
* Visual problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Type 1 diabetes followed in the department of Endocrinology, diabetology and nutrition (CHRU de Nancy)
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
success rate | 2 months
  score of the formation (80% correct answers)

SECONDARY OUTCOMES:
satisfaction measured by auto-questionnaire | 2 months
  calculation of total score of the answers on 6-point likert scale (minimum value = 0; maximum value = 100% , higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France